CLINICAL TRIAL: NCT00645060
Title: A Phase I Study of Yttrium-90 Labeled Humanized Anti-CEA M5A Antibody in Patients With CEA Producing Advanced Malignancies
Brief Title: Yttrium Y 90 DOTA Anti-CEA Monoclonal Antibody M5A in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05198; P30CA033572 (NIH); CHNMC-05198; CDR0000590300 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-03-26; First posted 2008-03-27 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Chromatography, High Pressure Liquid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Y-90-DOTA-M5A anti-CEA antibody (Experimental)
  Interventions: Other: high performance liquid chromatography; Other: pharmacological study; Procedure: radionuclide imaging; Procedure: single photon emission computed tomography; Radiation: yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A

INTERVENTIONS:
Other: high performance liquid chromatography — Performed on serial blood samples from 0 to 168 hours and daily X5 days 24 hour urine samples
Other: pharmacological study — Serial blood samples from 0 to 168 hours and daily X5 days 24 hour urine samples
Procedure: radionuclide imaging — 1-3 hours, 1 day, 2 days, 3-5 days and 6-7 days post Y-90 anti-CEA antibody infusion
Procedure: single photon emission computed tomography — 2 days and 3-5 days post antibody infusion
Radiation: yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A — Dose escalation from 12 mCi/m2 through 18 mCi/m2 increasing by 2 mCi/m2 with each escalation

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A, can find tumor cells and carry tumor-killing substances to them without harming normal cells. This may be an effective treatment for advanced cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish the maximum tolerated dose of yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A and describe the toxicities at each dose studied.
* To estimate radiation doses to whole body, normal organs, and tumor through serial nuclear imaging studies after intravenous infusion of the yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A.

OUTLINE: This is a dose-escalation study of yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A (MOAB M5A).

* Biodistribution: Patients receive indium In 111 radiolabeled anti-CEA MOAB M5A IV over 30 minutes. Patients undergo serial nuclear scans, single photon emission computed tomography (SPECT), and blood and urine sampling over 1 week to estimate absorbed radiation doses to tumor, normal organs (i.e., liver, lung, kidney, and bone marrow), and whole body.
* Treatment: No more than 2 weeks later, patients with adequate biodistribution receive yttrium Y 90 DOTA anti-CEA MOAB M5A IV over 30 minutes on day 1. Patients then undergo serial nuclear scans, SPECT, and blood and urine sampling over 1 week to estimate absorbed radiation doses to tumor, normal organs (i.e., liver, lung, kidney, and bone marrow), and whole body. Treatment repeats every 6-10 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Blood and urine samples are collected periodically for analysis of total activity by radiometric high performance liquid chromatography and to acquire data on antibody metabolism and pharmacokinetics.

After completion of study treatment, patients are followed every 3 months for up to 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor for which no standard or effective treatment is available

  * Patients who refuse an available standard but non-curative treatment may also be eligible
* Tumors must produce CEA as documented by either an elevated serum CEA above the upper limit of normal (ULN) or by immunohistochemical (IHC) methods

  * Positive CEA IHC stain is determined if more than 30% of the tumor cells have an intensity of 2+ or greater
* Measurable disease
* Estimated < 1/3 of liver involvement if tumor involves the liver
* No brain or leptomeningeal involvement with cancer

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* WBC ≥ 4,000/μL
* ANC ≥ 1,500/μL
* Platelet count ≥ 125,000/μL
* Creatinine ≤ 1.5 mg/dL and/or creatinine clearance > 60 mL/min
* Bilirubin ≤ 1.5 mg/dL
* ALT and AST ≤ 2 times ULN
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients currently being treated for severe infections or recovering from other intercurrent illnesses (such as poorly controlled diabetes or hypertension) are ineligible until recovery is deemed complete by the investigator
* Serum anti-antibody testing must be negative for human anti-humanized antibodies (if patient received prior monoclonal antibody)
* Serum HIV-negative
* Serum hepatitis B antigen- and hepatitis C antibody-negative

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior radiotherapy, immunotherapy, or chemotherapy (6 weeks for mitomycin C or nitrosoureas) and recovered
* Recovered from prior major surgery
* No prior radiotherapy to > 50% of bone marrow
* No other concurrent chemotherapy, radiotherapy, or immunotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10-09; Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 10 weeks after the beginning of the last cycle of treatment
Toxicity | From the date of the beginning of the first cycle of treatment to 10 weeks from the date of the beginning of the last cycle of treatment
Overall survival | From 3 months after treatment completion or until death
Progression-free survival | From 3 months after treatment completion until cancer progression or start of another treatment
Time to progression | 3 months and six months after treatment completion until cancer progression or start of another treatment
Pharmacokinetic and molecular studies | At 0, 1, 4-6, 12-24, 48, 72-120 and 144-168 hours after administration of the baseline imaging dose

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y. Wong, MD, Principal Investigator — City of Hope Comprehensive Cancer Center; Stephen I. Shibata, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States